CLINICAL TRIAL: NCT03515902
Title: The Effects of Mouthguard With Desensitizing Toothpaste in Reducing Dental Hypersensitivity in Swimmers : A Randomized Clinical Trial
Brief Title: The Effects of Mouthguard and Desensitizing Toothpaste in Reducing Dental Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Kemporn Kitsahawong, Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KKUHE612062
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-01

CONDITIONS: Dentine Hypersensitivity; Tooth Erosion
Keywords: Dentine Hypersensitivity; Toothpaste; Tooth erosion
MeSH Terms: conditions — Dentin Sensitivity; Tooth Erosion | interventions — Mouth Protectors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mouthguard (Experimental): Mouthguard arm is application of mouthguard while swimming
  Interventions: Device: mouthguard
- mouthguard with desensitizing toothpaste (Experimental): Mouthguard with desensitizing toothpaste arm is application of mouthguard with desensitizing toothpaste containing 8% arginine and calcium carbonate while swimming
  Interventions: Device: mouthguard with desensitizing toothpaste

INTERVENTIONS:
Device: mouthguard — mouthguard
  Arms: mouthguard
Device: mouthguard with desensitizing toothpaste — mouthguard with desensitizing toothpaste containing 8% arginine with calcium carbonate
  Arms: mouthguard with desensitizing toothpaste

SUMMARY:
Tooth hypersensitivity due to dental erosion is one of the most common problem related to swimming in improper pH chlorinated pools. Because the teeth are exposed to acidic water for a long time, which cause the loss of dental hard tissue. Tooth hypersensitivity can lead to a negative effect on daily life such as dietary selection, maintaining optimal dental hygiene and beauty aspects. It has been found that using mouthguard while swimming can prevent the teeth directly contact to chlorinated water, so it can protect tooth structure and decrease tooth hypersensitivity. Moreover, using mouthguard with viscous products can seal the gaps between mouthguard and teeth which can help to protect tooth structure and decrease dental hypersensitivity more effectively. At present, there are many desensitizing products such as toothpaste, mouthwash and chewing gum. Desensitizing toothpaste is the most common over-the-counter (OTC) materials in desensitizing. Many research has endorsed the properties of desensitizing toothpaste that can reduce tooth tissue loss and helps to reduce tooth hypersensitivity effectively. So it can be hypothesize that when use the combination of mouthguard with desensitizing toothpaste, it might have synergistic effect on reducing tooth hypersensitivity in swimmers.

DETAILED DESCRIPTION:
Tooth erosion is the loss of dental hard tissue due to acidic agents without bacteria involvement.

Mouthguard is a protective appliance use for covering the teeth and gums to prevent the teeth from acidic chlorinated water.

Desensitizing toothpaste is toothpaste containing 8 percent arginine and calcium carbonate that can reduce tooth demineralization and promote remineralization.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-25 years (age under 18 years must obtain consent from parents)
* Swimming at least 5 hours/week
* Having tooth hypersensitivity from erosion
* Can read or understand Thai language

Exclusion Criteria:

* History of allergic to toothpaste
* Having any tooth which will affect to the tightness of mouthguard
* Having fixed orthodontic appliance

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Tooth hypersensitivity changes after using mouthguard with/without desensitizing toothpaste | baseline,2,4 and 8 weeks
  * Tooth hypersensitivity changes will be measured by the mean difference of visual analog scale (VAS) score at baseline,2,4 and 8 weeks by using 2 clinical stimuli including tactile and cold stimulation. Each stimulation will be measured and separately recorded as follow :
    1.Tactile stimulation
  * The score range from 0 (no tooth hypersensitivity) to 100 (worst possibly tooth hypersensitivity)
  * The mean difference of tooth hypersensitivity from tactile stimulation at any time point will be analyzed.
    2. Cold stimulation
  * The score range from 0 (no tooth hypersensitivity) to 100 (worst possibly tooth hypersensitivity)
  * The mean difference of tooth hypersensitivity from cold stimulation at any time point will be analyzed.

SECONDARY OUTCOMES:
The attitude and satisfaction of using mouthguard with/without desensitizing toothpaste | 2,4 and 8 weeks
  * The attitude and satisfaction will be collected by a self-administered questionnaire and interview at 2,4 and 8 weeks
  * The score range from 0 (no satisfying) to 100 (most satisfying)
  * The mean score of satisfying at any time point will be analyzed.

OTHER OUTCOMES:
The quality of life after using mouthguard with/without desensitizing toothpaste | 8 weeks
  * The quality of life will be collected by interview at 8 weeks using oral impacts on daily performance (OIDP) questionnaire
  * The score range from 0 (no negative effect on quality of life) to 100 (worst negative effect on quality of life )
  * The mean score will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Kemporn Kitsahawong, DDS,MSc,PhD, Principal Investigator — Faculty of Dentistry, Khon Kaen University
Locations (1):
- Faculty of Dentistry , Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No